CLINICAL TRIAL: NCT02502981
Title: A Randomised Open Label, Blinded End Point Trial to Compare the Effects of Spironolactone With Chlortalidone on LV Mass in Stage 3 Chronic Kidney Disease (SPIRO-CKD)
Brief Title: Comparing the Effects of Spironolactone With Chlortalidone on LV Mass in Patients With CKD
Acronym: SPIRO-CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); University of Edinburgh (Other); University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr JN Townend, Professor of Cardiology, University Hospital Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP/12/8/29620
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Renal Insufficiency, Chronic; Cardio-Renal Syndrome
Keywords: CKD; left ventricle; aldosterone; spironolactone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardio-Renal Syndrome | interventions — Spironolactone; Mineralocorticoid Receptor Antagonists; Chlorthalidone; Sodium Chloride Symporter Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CKD stage 2 & 3 (Experimental): Patients with CKD stage 2 & 3 (eGFR 30-89ml/min/1.73m2) will be randomly assigned to receive either spironolactone or chlortalidone in a PROBE design.
  Subjects will undergo cardiac MRI, carotid femoral pulse wave velocity, 24 hour ambulatory blood pressure monitoring, blood tests for renal function and spot urine analysis for proteinuria (albumin:creatinine ratio) at baseline and after 40 weeks of allocated treatment. Additional blood tests for renal function and potassium level will be assessed at week 1,2,4,8 and 20.
  Interventions: Drug: Spironolactone; Drug: Chlortalidone

INTERVENTIONS:
Drug: Spironolactone — 25mg orally once a day for 40 weeks
  Other Names: Aldactone, Mineralocorticoid receptor antagonist
Drug: Chlortalidone — 25mg orally once a day for 40 weeks
  Other Names: Hygroton, Thalitone, Thiazide diuretic

SUMMARY:
In stage 3 chronic kidney disease (CKD) the risk of death due to cardiovascular causes is high and greatly exceeds the risk of progression to end stage renal failure. This high cardiovascular risk is predominantly due to sudden cardiac death and heart failure, manifestations of left ventricular hypertrophy and fibrosis. Aldosterone appears to play an important role in the causation of this myocardial disease both by direct inflammatory and fibrotic myocardial effects and via increased arterial stiffness due to hypertrophy, inflammation, and fibrosis within the media of large arteries. Levels of aldosterone are high in CKD despite sodium overload and treatment with angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) drugs due to the twin phenomena of aldosterone escape and breakthrough. In a previous British Heart Foundation funded study, Birmingham investigators showed that the addition of the mineralocorticoid receptor blocker (MRB) spironolactone to background therapy with ACE inhibitors or ARBs caused reductions in the prognostically important parameters of arterial stiffness and LV mass. Because spironolactone therapy was also associated with significant falls in arterial pressure it remains possible that these effects were mediated simply by blood pressure reduction. In this multi-centre, randomised controlled study, the effects of treatment with spironolactone on LV mass and arterial stiffness in patients with stage 3 CKD on established ACE or ARB therapy will be compared to those of chlortalidone, a control anti-hypertensive agent. Early stage chronic kidney disease is highly prevalent and new, cost effective treatment strategies are required to reduce cardiovascular risk. This study is designed to provide the rationale for a larger study of morbidity and mortality with MRB therapy in early stage CKD.

DETAILED DESCRIPTION:
Background

1. Chronic kidney disease and cardiovascular disease CKD is a major but poorly recognised and under-treated risk factor for cardiovascular disease. It can be categorised in to 5 stages according to GFR and the presence of markers of kidney damage. Stage 3 CKD, the subject of this proposal, is defined by a glomerular filtration rate (GFR) of 30-59 ml/min/1.73m2. There is a graded inverse relationship between cardiovascular risk and GFR which is independent of age, sex and other risk factors. There is also a graded association between albuminuria and cardiovascular risk and in patients with both low GFR and albuminuria, risk is increased with a multiplicative association. While the cardiovascular risk of end stage CKD is extreme, in public health terms the burden resides in early stage (CKD stages 1-3) disease, which is more prevalent affecting almost 1 in 7 of the entire population, including approximately 4% of those aged 40-59 and more than 40% of those over 70 years. Thus, CKD is a potentially important risk factor for cardiovascular disease in the general population. Although the risks of myocardial infarction and other manifestations of coronary artery disease are increased in CKD, there is a much greater increase in the incidence of heart failure and sudden cardiac death in stages 3-5. This is almost certainly a reflection of the very high prevalence of myocardial disease; left ventricular hypertrophy (LVH) often accompanied by magnetic resonance imaging evidence of fibrosis is present in over 30% of patients with stage 2 (GFR 60-89) and stage 3 CKD and in 80% of patients at the start of renal replacement therapy. To date, the only prospective trial to examine the prognostic benefit of drug therapy in this high risk group is the recently presented SHARP trial. This showed a reduction in occlusive vascular events associated with LDL lowering with simvastatin and ezetimibe. The Birmingham CRIB-2 study (see below) published in 2010 provided evidence that mineralocorticoid receptor blockade with spironolactone exerts beneficial effects on intermediate end points of strong prognostic value including LV mass and arterial stiffness. That work provides the basis for this application.

   Pathophysiology of myocardial and vascular disease in chronic kidney disease

   The main pathological features of cardiovascular disease in CKD are:
   1. Myocardial disease characterised by LVH and fibrosis accompanied by systolic and diastolic dysfunction.
   2. Arterial wall thickening, stiffening and calcification (arteriosclerosis).
   3. Coronary and peripheral artery atherosclerosis.

   Although there is no doubt that patients with CKD are subject to accelerated atherosclerosis the major pathological features of the cardiovascular system in CKD are myocardial disease (so called uraemic cardiomyopathy) and arterial stiffening due to arteriosclerosis. As kidney function declines, a range of abnormalities occur that may exert adverse effects upon the cardiovascular system. Hypertension, chronic anaemia, oxidative stress, inflammation and activation of the renin-angiotensin-aldosterone (RAAS) and sympathetic nervous systems all appear to contribute to the development of atherosclerosis, arteriosclerosis and myocardial hypertrophy and fibrosis.
2. Aldosterone and Cardiovascular Disease The fundamental role of the RAAS in cardiovascular disease is apparent from the results of many large ACE inhibitor trials showing mortality benefit in patients with chronic heart failure and in those with, or at high risk of, coronary artery disease. These beneficial effects have been attributed to prevention of the multiple adverse effects of angiotensin II. Strong evidence suggests that aldosterone may also be an important mediator of cardiac and vascular damage in many disease states. In trials involving patients with chronic heart failure and heart failure complicating myocardial infarction, the addition of the MRBs - spironolactone (RALES) or eplerenone (EPHESUS and EMPHASIS ) - to standard therapy including ACE inhibition reduced mortality by up to 30%. Primary aldosteronism is associated with a greater LV mass and higher risk of adverse cardiovascular events than control hypertensive populations and in patients after myocardial infarction, plasma aldosterone concentration even within the normal range predicts an adverse prognosis. More recently, a study of subjects undergoing coronary angiography confirmed an independent association of plasma aldosterone levels with total and cardiovascular mortality.

The mechanisms of action of aldosterone include upregulation of Angiotensin 1 receptors and direct effects on fibroblast collagen synthesis as well as decreased matrix metallo-proteinase secretion. An anti-fibrotic effect of MRB therapy may be of major importance. After myocardial infarction, circulating markers of collagen turnover and fibrosis were reduced by MRB therapy and in the RALES study myocardial collagen turnover was significantly reduced by spironolactone and the fall in the marker of this index was related to the mortality benefit. In CKD stages 2 and 3, data from CRIB-2 showed that spironolactone improves myocardial diastolic function and collagen turnover. .

Use of MRBs in Patients with CKD Although some doubt remains about whether ACE inhibitors and ARBs are superior to other blood pressure lowering drugs in slowing the progression of CKD, they may provide marginal extra benefit and are widely recommended in national and international guidelines. Conversely, the traditional approach by nephrologists to MRB drugs has been to avoid their use because of the risk of azotaemia and hyperkalaemia. There are both theoretical and empirical reasons why this avoidance may be incorrect. Firstly, CKD is characterised by an abnormal combination of chronic sodium overload and high (unsuppressed) levels of circulating aldosterone; the normal relationship between circulating volume and aldosterone secretion appears to be altered (aldosterone escape). Secondly, in a large proportion of patients with CKD on standard treatment with ACE inhibitors or ARBs, there is aldosterone 'breakthrough' so that aldosterone levels are high despite inhibition of the system by prevention of angiotensin II formation or inhibition of angiotensin receptors. Thus patients with CKD are exposed to high levels of aldosterone despite standard treatment. The only other common disease state in which high aldosterone production continues to occur in the face of sodium overload is chronic heart failure in which MRB therapy is of major prognostic benefit reducing both adverse cardiovascular events and total mortality.

There is also accumulating evidence to suggest that the addition of MRBs to ACE inhibitors in CKD might have beneficial effects by slowing the otherwise progressive decline in renal function. Animal experiments have shown that aldosterone can mediate renal injury and that MRBs such as eplerenone effectively reduce this. MRBs remain effective in low aldosterone models of CKD probably reflecting the importance of local (paracrine) aldosterone synthesis. In humans, small studies have suggested that the addition of MRBs to ACE inhibitors or ARB reduces proteinuria and may slow the progression of renal disease. Thus, the widespread use of MRBs in CKD has been advocated and has even been termed 'renal aspirin'. Until the publication of the CRIB-2 trial however, little attention had been paid to the potentially beneficial effects of MRB therapy on the cardiovascular system in patients with CKD.

The CRIB-2 trial The Effect of Spironolactone on Left Ventricular Mass and Aortic Stiffness in Early-Stage Chronic Kidney Disease; a Randomised Controlled Trial In a placebo controlled double blind trial, 112 patients (mean age 54 years) with stage 2 and 3 CKD with good blood pressure control on established treatment with ACE inhibitors or ARBs were treated in an active run-in phase with spironolactone 25 mg once daily for 4 weeks and then randomised to continue spironolactone or to receive a matching placebo for a total of 40 weeks. LV mass (cardiac magnetic resonance) and arterial stiffness (pulse wave velocity/analysis, aortic distensibility) were measured before run in and after 40 weeks of treatment. Compared with placebo, the use of spironolactone resulted in large reductions in LV mass and arterial stiffness (pulse wave velocity, augmentation index and aortic distensibility). This trial has been well received and widely publicised. In a recent review, Pitt stated that "we can be cautiously optimistic that use of an MRB in addition to an ACE inhibitor or an ARB will reduce the mortality and morbidity associated with CKD, as well as prevent its progression to end-stage renal disease with all of its health-care and health-cost consequences". Thus, this old and inexpensive drug has the potential to reduce adverse cardiovascular events and mortality in early stage CKD, a risk factor that is now screened for routinely in primary care by measurement of eGFR in the United Kingdom population. In the CRIB-2 trial, systolic blood pressure was significantly reduced; spironolactone is well recognised as an effective anti-hypertensive agent for patients with hypertension, even when this is resistant to other drugs. It is therefore necessary to determine whether the improvements in arterial stiffness and LV mass that occurred with spironolactone were mediated by this effect. Furthermore, before a large scale clinical trial of spironolactone can be contemplated, it is necessary to demonstrate that spironolactone can be used safely in a multi-centre trial design with local monitoring of renal function and serum potassium. This study will provide the pilot data on efficacy (independent of blood pressure) and safety that are necessary to undertake a definitive phase III trial of the role of spironolactone in reducing cardiovascular morbidity and mortality in patients with early stage CKD.

Recruitment and sample size

The trial started recruitment in June 2014, and aimed to recruit 350 patients over a 2 year period. The study was originally planned to be complete by February 2017. The rate of recruitment however was much slower than anticipated and it became evident by November 2015 that it would take a further 2 years to reach this target. This period of time was greater than funding allowed and the decision was taken to change the study design.

The initial design of the study was to use a co-primary end point of change in LV mass and change in pulse wave velocity. A sample size of 350 patients was planned to give 90% power to detect a difference in PWV with a p value of 0.025 and >90% power to detect a change in LV mass. When it became evident that was not achievable within the funded time frame the study was re-designed using the single end point of change in LV mass. With a p value of 0.05 and a power of 85%, it was calculated that 63 patients per group would be required. The sample size was calculated at 150 patients allowing for a 15% rate of missing data. This allowed a smaller sample size which was achievable within the funded time frame.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Chronic kidney disease stage 2 or 3 (eGFR 30-89 ml/min/1.73m2 by Modification of Diet in Renal Disease equation). eGFR must be within the last 12 months, on at least 2 occasions, at least 90 days apart.
* Well controlled blood pressure
* Established (>6 weeks) on treatment with ACE inhibitors or ARBs
* Not pregnant or breast feeding
* Males of childbearing age will be required to use medically approved contraception during and for 6 weeks following the last dose of study treatment.

Exclusion Criteria:

* Diabetes mellitus
* Clinical evidence of hypovolaemia
* Recent (< 6 months) acute myocardial infarction or other major adverse cardiovascular event (STEMI, NSTEMI, unstable angina, coronary revascularization, stroke, transient ischaemic attack)
* Known left ventricular systolic dysfunction ( ejection fraction <50%) or severe valvular heart disease
* Active malignant disease with a life expectancy of <5 years
* Previous hyperkalaemia (K+ >6.0 mmol/l) without precipitating cause
* Serum K+ >5.0 mmol/l at entry
* Serum sodium <130 mmol/l at entry
* Atrial fibrillation on screening ECG
* Use of a thiazide or loop diuretic in the 6 weeks prior to enrolment
* Pregnant or breastfeeding
* Known alcohol or drug abuse
* Active chronic diarrhea
* Recent active gout (within 3 months)
* Acute kidney injury in previous 3 months
* Documented Addison's disease
* On treatment with fludrocortisone, co-trimoxazole and / or lithium therapy
* Combination treatment with ACE inhibitor and ARB
* Office blood pressure <115 mmHg systolic or <50 mmHg diastolic
* Office blood pressure uncontrolled and requiring urgent non trial treatment in the opinion of the investigator
* Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-06; Primary Completion 2018-02 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change in LV mass measured by cardiac MRI | week 40

SECONDARY OUTCOMES:
Change in arterial stiffness measured by carotid-femoral pulse wave velocity | up to week 40
Change in serum potassium | up to week 40
  Potassium will be assessed at baseline, week 1,2,4,8,20 and week 40
Change in 24 hour ambulatory blood pressure | up to week 40
  Patients will wear an ambulatory monitor at week 0 and 40
Change in left ventricular systolic function as measured by Global longitudinal strain using MR tagging | up to week 40
  Global longitudinal strain (%) will be assessed at week 0 and 40
Change in renal function | up to week 40
  Estimated GFR will calculated using the Modification of Diet in Renal Disease equation at baseline, week 1,2,4,8,20 and week 40

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Slinn, Study Director — University of Birmingham
Locations (4):
- United Kingdom (4):
  - Departments of Cardiology & Nephrology University Hospital Birmingham, Birmingham, West Midlands
  - Cambridge Clinical Trials Unit, University of Cambridge and Addenbrooke's Hospital, Cambridge
  - University of Edinburgh: BHF Centre for Cardiovascular Science and Western General Hospital, Edinburgh
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Edwards NC, Ferro CJ, Townend JN, Steeds RP. Aortic distensibility and arterial-ventricular coupling in early chronic kidney disease: a pattern resembling heart failure with preserved ejection fraction. Heart. 2008 Aug;94(8):1038-43. doi: 10.1136/hrt.2007.137539. Epub 2008 Feb 28. PMID 18308865
- [Background] Edwards NC, Steeds RP, Stewart PM, Ferro CJ, Townend JN. Effect of spironolactone on left ventricular mass and aortic stiffness in early-stage chronic kidney disease: a randomized controlled trial. J Am Coll Cardiol. 2009 Aug 4;54(6):505-12. doi: 10.1016/j.jacc.2009.03.066. PMID 19643310
- [Background] Chue CD, Townend JN, Steeds RP, Ferro CJ. Arterial stiffness in chronic kidney disease: causes and consequences. Heart. 2010 Jun;96(11):817-23. doi: 10.1136/hrt.2009.184879. Epub 2010 Apr 20. PMID 20406771
- [Background] Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, Palensky J, Wittes J. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999 Sep 2;341(10):709-17. doi: 10.1056/NEJM199909023411001. PMID 10471456
- [Background] Brown NJ. Aldosterone and vascular inflammation. Hypertension. 2008 Feb;51(2):161-7. doi: 10.1161/HYPERTENSIONAHA.107.095489. Epub 2008 Jan 2. No abstract available. PMID 18172061
- [Background] Struthers AD. Aldosterone: cardiovascular assault. Am Heart J. 2002 Nov;144(5 Suppl):S2-7. doi: 10.1067/mhj.2002.129969. PMID 12422134
- [Background] Rocha R, Stier CT Jr, Kifor I, Ochoa-Maya MR, Rennke HG, Williams GH, Adler GK. Aldosterone: a mediator of myocardial necrosis and renal arteriopathy. Endocrinology. 2000 Oct;141(10):3871-8. doi: 10.1210/endo.141.10.7711. PMID 11014244
- [Background] Zannad F, Alla F, Dousset B, Perez A, Pitt B. Limitation of excessive extracellular matrix turnover may contribute to survival benefit of spironolactone therapy in patients with congestive heart failure: insights from the randomized aldactone evaluation study (RALES). Rales Investigators. Circulation. 2000 Nov 28;102(22):2700-6. doi: 10.1161/01.cir.102.22.2700. PMID 11094035
- [Background] Edwards NC, Ferro CJ, Kirkwood H, Chue CD, Young AA, Stewart PM, Steeds RP, Townend JN. Effect of spironolactone on left ventricular systolic and diastolic function in patients with early stage chronic kidney disease. Am J Cardiol. 2010 Nov 15;106(10):1505-11. doi: 10.1016/j.amjcard.2010.07.018. PMID 21059444
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, Safar ME, London GM. Impact of aortic stiffness on survival in end-stage renal disease. Circulation. 1999 May 11;99(18):2434-9. doi: 10.1161/01.cir.99.18.2434. PMID 10318666
- [Background] Matsumoto Y, Hamada M, Hiwada K. Aortic distensibility is closely related to the progression of left ventricular hypertrophy in patients receiving hemodialysis. Angiology. 2000 Nov;51(11):933-41. doi: 10.1177/000331970005101106. PMID 11103862
- [Background] Rahman M, Pressel S, Davis BR, Nwachuku C, Wright JT Jr, Whelton PK, Barzilay J, Batuman V, Eckfeldt JH, Farber M, Henriquez M, Kopyt N, Louis GT, Saklayen M, Stanford C, Walworth C, Ward H, Wiegmann T. Renal outcomes in high-risk hypertensive patients treated with an angiotensin-converting enzyme inhibitor or a calcium channel blocker vs a diuretic: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Arch Intern Med. 2005 Apr 25;165(8):936-46. doi: 10.1001/archinte.165.8.936. PMID 15851647
- [Background] Smith DH, Neutel JM, Lacourciere Y, Kempthorne-Rawson J. Prospective, randomized, open-label, blinded-endpoint (PROBE) designed trials yield the same results as double-blind, placebo-controlled trials with respect to ABPM measurements. J Hypertens. 2003 Jul;21(7):1291-8. doi: 10.1097/00004872-200307000-00016. PMID 12817175
- [Background] Mark PB, Johnston N, Groenning BA, Foster JE, Blyth KG, Martin TN, Steedman T, Dargie HJ, Jardine AG. Redefinition of uremic cardiomyopathy by contrast-enhanced cardiac magnetic resonance imaging. Kidney Int. 2006 May;69(10):1839-45. doi: 10.1038/sj.ki.5000249. PMID 16508657
- [Result] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577